CLINICAL TRIAL: NCT00115934
Title: Trial of Right Ventricular Versus Modified Blalock-Taussig Shunt in Infants With Single Ventricle Defect Undergoing Staged Reconstruction (A Trial Conducted by the Pediatric Heart Network)
Brief Title: Comparison of Two Types of Shunts in Infants With Single Ventricle Defect Undergoing Staged Reconstruction--Pediatric Heart Network
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carelon Research (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); Pediatric Heart Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 194; U01HL068270 (NIH); U01HL068269 (NIH); U01HL068279 (NIH); U01HL068281 (NIH); U01HL068285 (NIH); U01HL068288 (NIH); U01HL068290 (NIH); U01HL068292 (NIH)
Record Dates: First submitted 2005-06-26; First posted 2005-06-27 (Estimated); Results first posted 2011-06-27 (Estimated); Last update posted 2025-03-11 (Actual); Status verified 2013-08

CONDITIONS: Heart Defects, Congenital
MeSH Terms: conditions — Heart Defects, Congenital | interventions — Blalock-Taussig Procedure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MBTS (Active Comparator): Blalock-Taussig pulmonary artery shunt
  Interventions: Procedure: Blalock-Taussig pulmonary artery shunt
- RVPAS (Active Comparator): Right ventricular to pulmonary artery shunt
  Interventions: Procedure: Right ventricular to pulmonary artery shunt

INTERVENTIONS:
Procedure: Blalock-Taussig pulmonary artery shunt — Performed at stage I palliative surgery for babies born with HLHS
  Other Names: MBTS procedure
  Arms: MBTS
Procedure: Right ventricular to pulmonary artery shunt — Performed at stage I palliative surgery for babies born with HLHS
  Other Names: RV to PA or Sano procedure
  Arms: RVPAS

SUMMARY:
This trial will evaluate the efficacy and safety of the modified Blalock-Taussig shunt (MBTS) compared to the right ventricle to pulmonary artery (RV-to-PA) shunt; compare the effect of the MBTS to that of the RV-to-PA shunt on the incidence of death or cardiac transplantation at 12 months post randomization; and compare the effect of the two shunts on intensive care unit (ICU) morbidity, unintended cardiovascular interventional procedures, right ventricular function, tricuspid valve regurgitation, pulmonary artery growth, and neurodevelopmental outcome.

DETAILED DESCRIPTION:
BACKGROUND:

Hypoplastic left heart syndrome (HLHS) and related single right ventricle anomalies are the highest risk congenital cardiovascular malformations. Surgical repair begins with the Norwood procedure during the newborn period, a stage II procedure at 4 to 6 months of age, and Fontan procedure at 18 to 36 months. The Norwood procedure remains one of the highest risk procedures in congenital heart surgery. A few small nonrandomized studies of a novel approach to the Norwood procedure have reported improved outcomes. This new approach uses a RV-to-PA shunt to provide pulmonary blood flow rather than the standard MBTS. This multi-center, randomized clinical trial will evaluate early and intermediate-term outcomes for patients undergoing a Norwood procedure with either the RV-to-PA shunt or the MBTS.

This study has been approved by the Institutional Review/Research Ethics Boards of all participating clinical centers:

Hospital for Sick Children, Toronto, Canada

Children's Hospital Boston, Boston, MA

Columbia College of Physicians and Surgeons, New York, NY

Children's Hospital of Philadelphia, Philadelphia, PA

Duke University Medical Center, Durham, NC

Brody School of Medicine at East Carolina University, Greenville, NC

Wake Forest Baptist Medical Center, Winston Salem, NC

Medical University of South Carolina, Charleston, SC

Children's Hospital of Wisconsin, Milwaukee, WI

University of Michigan, Ann Arbor, MI

Cincinnati Children's Hospital Medical Center, Cincinnati, OH

Children's Hospital of Los Angeles, Los Angeles, CA

Egleston Children's Hospital, Emory University, Atlanta, GA

Congenital Heart Institute of Florida, University of South Florida, St. Petersburg, FL

Alfred I. duPont Hospital for Children, Wilmington, DE

DESIGN NARRATIVE:

This is a prospective, randomized clinical trial of the RV-to-PA shunt versus MBTS in patients undergoing a Norwood procedure.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hypoplastic left heart syndrome or related single, morphologic right ventricle anomaly
* Planned Norwood procedure
* Informed consent of parent(s) or legal guardian

Exclusion Criteria:

* Single, morphologic left ventricle anomaly
* Preoperative identification of anatomy rendering either an MBTS or an RV-to-PA shunt technically impossible
* Any major congenital abnormality (i.e., congenital diaphragmatic hernia, tracheoesophageal fistula) or acquired extra-cardiac disorder (e.g., meconium aspiration with need for high frequency ventilation, persistent renal failure requiring dialysis) that, in the opinion of the investigator, could independently affect the likelihood of the subject meeting the primary endpoint

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 555 (Actual)
Dates: Start 2005-05; Primary Completion 2009-09 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julie E Miller, MPH, Principal Investigator — New England Research Institutes, Watertown, MA
Locations (13):
- United States (12):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Cardiac Surgical Associates, St. Petersburg, Florida
  - Children's Healthcare of Atlanta at Egleston, Atlanta, Georgia
  - Children's Hospital Boston, Boston, Massachusetts
  - University of Michigan Health System/Mott Hospital, Ann Arbor, Michigan
  - Columbia College of Physicians and Surgeons, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Background] Ohye RG, Gaynor JW, Ghanayem NS, Goldberg CS, Laussen PC, Frommelt PC, Newburger JW, Pearson GD, Tabbutt S, Wernovsky G, Wruck LM, Atz AM, Colan SD, Jaggers J, McCrindle BW, Prakash A, Puchalski MD, Sleeper LA, Stylianou MP, Mahony L; Pediatric Heart Network Investigators. Design and rationale of a randomized trial comparing the Blalock-Taussig and right ventricle-pulmonary artery shunts in the Norwood procedure. J Thorac Cardiovasc Surg. 2008 Oct;136(4):968-75. doi: 10.1016/j.jtcvs.2008.01.013. Epub 2008 May 19. PMID 18954638
- [Result] Johnson JN, Ansong AK, Li JS, Xu M, Gorentz J, Hehir DA, del Castillo SL, Lai WW, Uzark K, Pasquali SK. Celiac artery flow pattern in infants with single right ventricle following the Norwood procedure with a modified Blalock-Taussig or right ventricle to pulmonary artery shunt. Pediatr Cardiol. 2011 Apr;32(4):479-86. doi: 10.1007/s00246-011-9906-y. Epub 2011 Feb 18. PMID 21331516
- [Result] Virzi L, Pemberton V, Ohye RG, Tabbutt S, Lu M, Atz TC, Barnard T, Dunbar-Masterson C, Ghanayem NS, Jacobs JP, Lambert LM, Lewis A, Pike N, Pizarro C, Radojewski E, Teitel D, Xu M, Pearson GD. Reporting adverse events in a surgical trial for complex congenital heart disease: the Pediatric Heart Network experience. J Thorac Cardiovasc Surg. 2011 Sep;142(3):531-7. doi: 10.1016/j.jtcvs.2010.11.052. Epub 2011 Mar 12. PMID 21397260
- [Result] Atz AM, Travison TG, Williams IA, Pearson GD, Laussen PC, Mahle WT, Cook AL, Kirsh JA, Sklansky M, Khaikin S, Goldberg C, Frommelt M, Krawczeski C, Puchalski MD, Jacobs JP, Baffa JM, Rychik J, Ohye RG; Pediatric Heart Network Investigators. Prenatal diagnosis and risk factors for preoperative death in neonates with single right ventricle and systemic outflow obstruction: screening data from the Pediatric Heart Network Single Ventricle Reconstruction Trial( *). J Thorac Cardiovasc Surg. 2010 Dec;140(6):1245-50. doi: 10.1016/j.jtcvs.2010.05.022. Epub 2010 Jun 18. PMID 20561642
- [Result] Ohye RG, Sleeper LA, Mahony L, Newburger JW, Pearson GD, Lu M, Goldberg CS, Tabbutt S, Frommelt PC, Ghanayem NS, Laussen PC, Rhodes JF, Lewis AB, Mital S, Ravishankar C, Williams IA, Dunbar-Masterson C, Atz AM, Colan S, Minich LL, Pizarro C, Kanter KR, Jaggers J, Jacobs JP, Krawczeski CD, Pike N, McCrindle BW, Virzi L, Gaynor JW; Pediatric Heart Network Investigators. Comparison of shunt types in the Norwood procedure for single-ventricle lesions. N Engl J Med. 2010 May 27;362(21):1980-92. doi: 10.1056/NEJMoa0912461. PMID 20505177
- [Result] Ohye RG, Devaney EJ, Hirsch JC, Bove EL. The modified Blalock-Taussig shunt versus the right ventricle-to-pulmonary artery conduit for the Norwood procedure. Pediatr Cardiol. 2007 Mar-Apr;28(2):122-5. doi: 10.1007/s00246-006-1449-2. Epub 2007 Feb 16. PMID 17308942
- [Derived] Mahle WT, Keesari R, Trachtenberg F, Newburger JW, Lim H, Edelson J, Jeewa A, Lal A, Kindel SJ, Burns KM, Lang S, Bainton J, Carboni M, Villa CR, Richmond M, Henderson H, Menteer J, Pizarro C, Goldberg CS. School age and adolescent heart failure following the Norwood procedure. J Heart Lung Transplant. 2024 Mar;43(3):453-460. doi: 10.1016/j.healun.2023.10.012. Epub 2023 Oct 20. PMID 37866470
- [Derived] Dolgner SJ, Tjoeng YL, Chan T. Analysis of the Single Ventricle Reconstruction Trial Using Restricted Mean Survival Time and Shunt Type Received. J Am Heart Assoc. 2022 Sep 20;11(18):e025978. doi: 10.1161/JAHA.122.025978. Epub 2022 Sep 8. No abstract available. PMID 36073629
- [Derived] Miller TA, Ghanayem NS, Newburger JW, McCrindle BW, Hu C, DeWitt AG, Cnota JF, Tractenberg FL, Pemberton VL, Wolf MJ, Votava-Smith JK, Fifer CG, Lambert LM, Shah A, Graham EM, Pizarro C, Jacobs JP, Miller SG, Minich LL; Pediatric Heart Network Investigators. Gestational Age, Birth Weight, and Outcomes Six Years After the Norwood Procedure. Pediatrics. 2019 May;143(5):e20182577. doi: 10.1542/peds.2018-2577. Epub 2019 Apr 12. PMID 30979811
- [Derived] Frommelt PC, Hu C, Trachtenberg F, Baffa JM, Boruta RJ, Chowdhury S, Cnota JF, Dragulescu A, Levine JC, Lu J, Mercer-Rosa L, Miller TA, Shah A, Slesnick TC, Stapleton G, Stelter J, Wong P, Newburger JW. Impact of Initial Shunt Type on Echocardiographic Indices in Children After Single Right Ventricle Palliations. Circ Cardiovasc Imaging. 2019 Feb;12(2):e007865. doi: 10.1161/CIRCIMAGING.118.007865. PMID 30755054
- [Derived] Mahle WT, Hu C, Trachtenberg F, Menteer J, Kindel SJ, Dipchand AI, Richmond ME, Daly KP, Henderson HT, Lin KY, McCulloch M, Lal AK, Schumacher KR, Jacobs JP, Atz AM, Villa CR, Burns KM, Newburger JW; Pediatric Heart Network Investigators. Heart failure after the Norwood procedure: An analysis of the Single Ventricle Reconstruction Trial. J Heart Lung Transplant. 2018 Jul;37(7):879-885. doi: 10.1016/j.healun.2018.02.009. Epub 2018 Feb 16. PMID 29571602
- [Derived] Newburger JW, Sleeper LA, Gaynor JW, Hollenbeck-Pringle D, Frommelt PC, Li JS, Mahle WT, Williams IA, Atz AM, Burns KM, Chen S, Cnota J, Dunbar-Masterson C, Ghanayem NS, Goldberg CS, Jacobs JP, Lewis AB, Mital S, Pizarro C, Eckhauser A, Stark P, Ohye RG; Pediatric Heart Network Investigators. Transplant-Free Survival and Interventions at 6 Years in the SVR Trial. Circulation. 2018 May 22;137(21):2246-2253. doi: 10.1161/CIRCULATIONAHA.117.029375. Epub 2018 Feb 1. PMID 29437119
- [Derived] Bucholz EM, Sleeper LA, Newburger JW. Neighborhood Socioeconomic Status and Outcomes Following the Norwood Procedure: An Analysis of the Pediatric Heart Network Single Ventricle Reconstruction Trial Public Data Set. J Am Heart Assoc. 2018 Feb 2;7(3):e007065. doi: 10.1161/JAHA.117.007065. PMID 29420218
- [Derived] Ramroop R, Manase G, Lu D, Manase D, Chen S, Kim R, Lee T, Mahle WT, McHugh K, Mitchell M, Tristani-Firouzi M, Wechsler SB, Wilder NS, Zak V, Lafreniere-Roula M, Newburger JW, Gaynor JW, Russell MW, Mital S. Adrenergic receptor genotypes influence postoperative outcomes in infants in the Single-Ventricle Reconstruction Trial. J Thorac Cardiovasc Surg. 2017 Nov;154(5):1703-1710.e3. doi: 10.1016/j.jtcvs.2017.06.041. Epub 2017 Jun 24. PMID 28734628
- [Derived] Meza JM, Hickey EJ, Blackstone EH, Jaquiss RDB, Anderson BR, Williams WG, Cai S, Van Arsdell GS, Karamlou T, McCrindle BW. The Optimal Timing of Stage 2 Palliation for Hypoplastic Left Heart Syndrome: An Analysis of the Pediatric Heart Network Single Ventricle Reconstruction Trial Public Data Set. Circulation. 2017 Oct 31;136(18):1737-1748. doi: 10.1161/CIRCULATIONAHA.117.028481. Epub 2017 Jul 7. PMID 28687711
- [Derived] Chowdhury SM, Graham EM, Atz AM, Bradley SM, Kavarana MN, Butts RJ. Validation of a Simple Score to Determine Risk of Hospital Mortality After the Norwood Procedure. Semin Thorac Cardiovasc Surg. 2016 Summer;28(2):425-433. doi: 10.1053/j.semtcvs.2016.04.004. Epub 2016 Apr 19. PMID 28043455
- [Derived] Burch PT, Ravishankar C, Newburger JW, Lambert LM, Pemberton VL, Granger S, Floh AA, Anderson JB, Hill GD, Hill KD, Oster ME, Lewis AB, Schumacher KR, Zyblewski SC, Davies RR, Jacobs JP, Lai WW, Minich LL; Pediatric Heart Network Investigators. Assessment of Growth 6 Years after the Norwood Procedure. J Pediatr. 2017 Jan;180:270-274.e6. doi: 10.1016/j.jpeds.2016.09.048. Epub 2016 Nov 14. PMID 27855999
- [Derived] Plummer ST, Hornik CP, Baker H, Fleming GA, Foerster S, Ferguson ME, Glatz AC, Hirsch R, Jacobs JP, Lee KJ, Lewis AB, Li JS, Martin M, Porras D, Radtke WA, Rhodes JF, Vincent JA, Zampi JD, Hill KD. Maladaptive aortic properties after the Norwood procedure: An angiographic analysis of the Pediatric Heart Network Single Ventricle Reconstruction Trial. J Thorac Cardiovasc Surg. 2016 Aug;152(2):471-479.e3. doi: 10.1016/j.jtcvs.2016.03.091. Epub 2016 Apr 14. PMID 27167022
- [Derived] Yilmaz B, Narayan HK, Wilpers A, Wiess C, Fifer WP, Williams IA. Electrocardiographic intervals in foetuses with CHD. Cardiol Young. 2016 Jan;26(1):84-9. doi: 10.1017/S1047951114002686. Epub 2015 Jan 20. PMID 25599806
- [Derived] Frommelt PC, Gerstenberger E, Cnota JF, Cohen MS, Gorentz J, Hill KD, John JB, Levine JC, Lu J, Mahle WT, McCandless RT, Mertens L, Pearson GD, Spencer C, Thacker D, Williams IA, Wong PC, Newburger JW; Pediatric Heart Network Investigators. Impact of initial shunt type on cardiac size and function in children with single right ventricle anomalies before the Fontan procedure: the single ventricle reconstruction extension trial. J Am Coll Cardiol. 2014 Nov 11;64(19):2026-35. doi: 10.1016/j.jacc.2014.08.033. Epub 2014 Nov 3. PMID 25440099
- [Derived] Burch PT, Gerstenberger E, Ravishankar C, Hehir DA, Davies RR, Colan SD, Sleeper LA, Newburger JW, Clabby ML, Williams IA, Li JS, Uzark K, Cooper DS, Lambert LM, Pemberton VL, Pike NA, Anderson JB, Dunbar-Masterson C, Khaikin S, Zyblewski SC, Minich LL; Pediatric Heart Network Investigators. Longitudinal assessment of growth in hypoplastic left heart syndrome: results from the single ventricle reconstruction trial. J Am Heart Assoc. 2014 Jun 23;3(3):e000079. doi: 10.1161/JAHA.114.000079. PMID 24958780
- [Derived] Goldberg CS, Lu M, Sleeper LA, Mahle WT, Gaynor JW, Williams IA, Mussatto KA, Ohye RG, Graham EM, Frank DU, Jacobs JP, Krawczeski C, Lambert L, Lewis A, Pemberton VL, Sananes R, Sood E, Wechsler SB, Bellinger DC, Newburger JW; Pediatric Heart Network Investigators. Factors associated with neurodevelopment for children with single ventricle lesions. J Pediatr. 2014 Sep;165(3):490-496.e8. doi: 10.1016/j.jpeds.2014.05.019. Epub 2014 Jun 19. PMID 24952712
- [Derived] Newburger JW, Sleeper LA, Frommelt PC, Pearson GD, Mahle WT, Chen S, Dunbar-Masterson C, Mital S, Williams IA, Ghanayem NS, Goldberg CS, Jacobs JP, Krawczeski CD, Lewis AB, Pasquali SK, Pizarro C, Gruber PJ, Atz AM, Khaikin S, Gaynor JW, Ohye RG; Pediatric Heart Network Investigators. Transplantation-free survival and interventions at 3 years in the single ventricle reconstruction trial. Circulation. 2014 May 20;129(20):2013-20. doi: 10.1161/CIRCULATIONAHA.113.006191. Epub 2014 Apr 4. PMID 24705119
- [Derived] Lambert LM, Pike NA, Medoff-Cooper B, Zak V, Pemberton VL, Young-Borkowski L, Clabby ML, Nelson KN, Ohye RG, Trainor B, Uzark K, Rudd N, Bannister L, Korsin R, Cooper DS, Pizarro C, Zyblewski SC, Bartle BH, Williams RV; Pediatric Heart Network Investigators. Variation in feeding practices following the Norwood procedure. J Pediatr. 2014 Feb;164(2):237-42.e1. doi: 10.1016/j.jpeds.2013.09.042. Epub 2013 Nov 6. PMID 24210923
- [Derived] Marx GR, Shirali G, Levine JC, Guey LT, Cnota JF, Baffa JM, Border WL, Colan S, Ensing G, Friedberg MK, Goldberg DJ, Idriss SF, John JB, Lai WW, Lu M, Menon SC, Ohye RG, Saudek D, Wong PC, Pearson GD; Pediatric Heart Network Investigators. Multicenter study comparing shunt type in the norwood procedure for single-ventricle lesions: three-dimensional echocardiographic analysis. Circ Cardiovasc Imaging. 2013 Nov;6(6):934-42. doi: 10.1161/CIRCIMAGING.113.000304. Epub 2013 Oct 4. PMID 24097422
- [Derived] Schwartz SM, Lu M, Ohye RG, Hill KD, Atz AM, Naim MY, Williams IA, Goldberg CS, Lewis A, Pigula F, Manning P, Pizarro C, Chai P, McCandless R, Dunbar-Masterson C, Kaltman JR, Kanter K, Sleeper LA, Schonbeck JV, Ghanayem N; Pediatric Heart Network Investigators. Risk factors for prolonged length of stay after the stage 2 procedure in the single-ventricle reconstruction trial. J Thorac Cardiovasc Surg. 2014 Jun;147(6):1791-8, 1798.e1-4. doi: 10.1016/j.jtcvs.2013.07.063. Epub 2013 Sep 24. PMID 24075564
- [Derived] Hill KD, Rhodes JF, Aiyagari R, Baker GH, Bergersen L, Chai PJ, Fleming GA, Fudge JC, Gillespie MJ, Gray RG, Hirsch R, Lee KJ, Li JS, Ohye RG, Oster ME, Pasquali SK, Pelech AN, Radtke WA, Takao CM, Vincent JA, Hornik CP. Intervention for recoarctation in the single ventricle reconstruction trial: incidence, risk, and outcomes. Circulation. 2013 Aug 27;128(9):954-61. doi: 10.1161/CIRCULATIONAHA.112.000488. Epub 2013 Jul 17. PMID 23864006
- [Derived] Williams IA, Fifer C, Jaeggi E, Levine JC, Michelfelder EC, Szwast AL. The association of fetal cerebrovascular resistance with early neurodevelopment in single ventricle congenital heart disease. Am Heart J. 2013 Apr;165(4):544-550.e1. doi: 10.1016/j.ahj.2012.11.013. Epub 2013 Feb 13. PMID 23537971
- [Derived] Bacha E, del Nido P. Introduction to the Single Ventricle Reconstruction trial. J Thorac Cardiovasc Surg. 2012 Oct;144(4):880-1. doi: 10.1016/j.jtcvs.2012.08.031. No abstract available. PMID 22980631
- [Derived] Ohye RG, Schonbeck JV, Eghtesady P, Laussen PC, Pizarro C, Shrader P, Frank DU, Graham EM, Hill KD, Jacobs JP, Kanter KR, Kirsh JA, Lambert LM, Lewis AB, Ravishankar C, Tweddell JS, Williams IA, Pearson GD; Pediatric Heart Network Investigators. Cause, timing, and location of death in the Single Ventricle Reconstruction trial. J Thorac Cardiovasc Surg. 2012 Oct;144(4):907-14. doi: 10.1016/j.jtcvs.2012.04.028. Epub 2012 Aug 15. PMID 22901498
- [Derived] Ghanayem NS, Allen KR, Tabbutt S, Atz AM, Clabby ML, Cooper DS, Eghtesady P, Frommelt PC, Gruber PJ, Hill KD, Kaltman JR, Laussen PC, Lewis AB, Lurito KJ, Minich LL, Ohye RG, Schonbeck JV, Schwartz SM, Singh RK, Goldberg CS; Pediatric Heart Network Investigators. Interstage mortality after the Norwood procedure: Results of the multicenter Single Ventricle Reconstruction trial. J Thorac Cardiovasc Surg. 2012 Oct;144(4):896-906. doi: 10.1016/j.jtcvs.2012.05.020. Epub 2012 Jul 11. PMID 22795436
- [Derived] Tabbutt S, Ghanayem N, Ravishankar C, Sleeper LA, Cooper DS, Frank DU, Lu M, Pizarro C, Frommelt P, Goldberg CS, Graham EM, Krawczeski CD, Lai WW, Lewis A, Kirsh JA, Mahony L, Ohye RG, Simsic J, Lodge AJ, Spurrier E, Stylianou M, Laussen P; Pediatric Heart Network Investigators. Risk factors for hospital morbidity and mortality after the Norwood procedure: A report from the Pediatric Heart Network Single Ventricle Reconstruction trial. J Thorac Cardiovasc Surg. 2012 Oct;144(4):882-95. doi: 10.1016/j.jtcvs.2012.05.019. Epub 2012 Jun 15. PMID 22704284
- [Derived] Pasquali SK, Ohye RG, Lu M, Kaltman J, Caldarone CA, Pizarro C, Dunbar-Masterson C, Gaynor JW, Jacobs JP, Kaza AK, Newburger J, Rhodes JF, Scheurer M, Silver E, Sleeper LA, Tabbutt S, Tweddell J, Uzark K, Wells W, Mahle WT, Pearson GD; Pediatric Heart Network Investigators. Variation in perioperative care across centers for infants undergoing the Norwood procedure. J Thorac Cardiovasc Surg. 2012 Oct;144(4):915-21. doi: 10.1016/j.jtcvs.2012.05.021. Epub 2012 Jun 12. PMID 22698562
- [Derived] Frommelt PC, Guey LT, Minich LL, Bhat M, Bradley TJ, Colan SD, Ensing G, Gorentz J, Heydarian H, John JB, Lai WW, Levine JC, Mahle WT, Miller SG, Ohye RG, Pearson GD, Shirali GS, Wong PC, Cohen MS; Pediatric Heart Network Investigators. Does initial shunt type for the Norwood procedure affect echocardiographic measures of cardiac size and function during infancy?: the Single Vventricle Reconstruction trial. Circulation. 2012 May 29;125(21):2630-8. doi: 10.1161/CIRCULATIONAHA.111.072694. Epub 2012 Apr 21. PMID 22523314
- [Derived] Newburger JW, Sleeper LA, Bellinger DC, Goldberg CS, Tabbutt S, Lu M, Mussatto KA, Williams IA, Gustafson KE, Mital S, Pike N, Sood E, Mahle WT, Cooper DS, Dunbar-Masterson C, Krawczeski CD, Lewis A, Menon SC, Pemberton VL, Ravishankar C, Atz TW, Ohye RG, Gaynor JW; Pediatric Heart Network Investigators. Early developmental outcome in children with hypoplastic left heart syndrome and related anomalies: the single ventricle reconstruction trial. Circulation. 2012 May 1;125(17):2081-91. doi: 10.1161/CIRCULATIONAHA.111.064113. Epub 2012 Mar 28. PMID 22456475
- [Derived] Tweddell JS, Sleeper LA, Ohye RG, Williams IA, Mahony L, Pizarro C, Pemberton VL, Frommelt PC, Bradley SM, Cnota JF, Hirsch J, Kirshbom PM, Li JS, Pike N, Puchalski M, Ravishankar C, Jacobs JP, Laussen PC, McCrindle BW; Pediatric Heart Network Investigators. Intermediate-term mortality and cardiac transplantation in infants with single-ventricle lesions: risk factors and their interaction with shunt type. J Thorac Cardiovasc Surg. 2012 Jul;144(1):152-9. doi: 10.1016/j.jtcvs.2012.01.016. Epub 2012 Feb 15. PMID 22341427

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects undergoing a Norwood were randomized to MBTS or RVPAS at 15 North American centers.
Pre-assignment Details: There were no pre-assignment requirements beyond the initial screening criteria.
Period: Overall Study
Arm/Group | MBTS | RVPAS
Started | 279 (279 randomized to MBTS, but 3 did not have a Norwood surgery; one was withdrawn-with limited data.) | 276 (276 randomized to RVPAS, but 2 did not have a Norwood surgery and were excluded from analyses.)
Completed | 275 | 274
Not Completed | 4 | 2
Not completed — Lost to Follow-up | 1 | 0
Not completed — Did not receive intervention | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MBTS | RVPAS | Total
Number analyzed (Participants) | 275 | 274 | 549
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 275 | 274 | 549
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: days] | 5.1 (4.1) | 5.0 (4.0) | 5.1 (4.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 107 | 102 | 209
  Male | 168 | 172 | 340
Region of Enrollment [Number; unit: participants]
  United States | 268 | 266 | 534
  Canada | 7 | 8 | 15

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients Who Died or Received a Heart Transplant
Description: The primary outcome was the proportion of patients who died or had cardiac transplantation 12 months after randomization.
Time Frame: Measured at 12 months
Population: 555 subjects were enrolled in the study; 5 of these subjects were excluded from analyses because a Norwood procedure was not performed; 1 subject was excluded because the subject withdrew before the 12-month follow-up, 12-month status was unknown. The data were analyzed on an intention to treat basis, subjects were analyzed as randomized.
Measure: Number; unit: Participants
Arm/Group | MBTS | RVPAS
Number analyzed (Participants) | 275 | 274
Participants | 100 | 72
Statistical Analysis 1: Comparison: MBTS vs RVPAS; The original sample size of 456 was based on 85% power, with a two-sided, two sample test of proportions (anticipating 28% MBTS subjects with events, 16% RVPAS subjects with events), and an alpha of 0.05. The critical p-value was 0.044 because four interim analyses were performed. The target trial size was increased from 466 to 554 to account for crossovers. The stopping boundary was crossed at the 4th interim look; however, the trial was not halted, because all subjects were enrolled; Test type: Superiority or Other; p = 0.013, Fisher Exact; Risk Difference (RD) = -10.1, 95% CI [-17.8 to -2.4] — The risk difference is defined as the percent of subjects with events in the RVPAS group minus the percent of subjects with events in the MBTS group

2. Secondary Outcome: Proportion of Deaths or Heart Transplants Over Time From Randomization to the End of the Trial
Description: This secondary outcome was the proportion of deaths or cardiac transplantation over time from randomization to the end of the trial.
Time Frame: From Randomization to the End of the Trial, an average of 32 months
Measure: Number; unit: Participants
Arm/Group | MBTS | RVPAS
Number analyzed (Participants) | 275 | 274
Participants | 107 | 88
Statistical Analysis 1: Comparison: MBTS vs RVPAS; Test type: Superiority or Other; p = 0.06, Log Rank

3. Secondary Outcome: Echocardiographic Measures of Heart Size and Function: Right Ventricle (RV) End-diastolic Volume Indexed to Body Surface Area (BSA)
Description: Right ventricular end-diastolic volume indexed to BSA^1.3. Echocardiograms were performed at time points relative to the two palliative surgeries (post-Norwood and pre-Stage II) as well as at the specific time point of 14 months of age.
Time Frame: Measured post-Norwood, an average of 17 days post-Norwood
Population: 241 and 239 patients remained in the MBTS and RVPAS groups at the time of the post-Norwood echo. Of these, some patients did not have acceptable echos or measures were not able to be obtained to calculate the volumes.
Measure: Median (Inter-Quartile Range); unit: ml/m^2.6
Arm/Group | MBTS | RVPAS
Number analyzed (Participants) | 173 | 194
ml/m^2.6 | 91.2 [76.3 to 108.1] | 86.5 [73.8 to 104.3]
Statistical Analysis 1: Comparison: MBTS vs RVPAS; Test type: Superiority or Other; p = 0.09, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Echocardiographic Measures of Heart Size and Function: RV End-diastolic Volume Indexed to BSA
Description: as for outcome 3
Time Frame: Measured pre-stage II surgery, an average of 15 days pre-stage II surgery
Population: 181 and 214 patients remained in the MBTS and RVPAS groups at the time of the pre-Stage II echo. Of these, some patients did not have acceptable echos or not all measures were able to be obtained to calculate the volumes.
Measure: Median (Inter-Quartile Range); unit: ml/m^2.6
Arm/Group | MBTS | RVPAS
Number analyzed (Participants) | 127 | 151
ml/m^2.6 | 113.4 [94.1 to 138.6] | 105.2 [86.8 to 125.3]
Statistical Analysis 1: Comparison: MBTS vs RVPAS; Test type: Superiority or Other; p = 0.009, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Echocardiographic Measures of Heart Size and Function: RV End-diastolic Volume Indexed to BSA
Description: as for outcome 3
Time Frame: Measured at 14 months of age
Population: 184 and 179 patients remained in the MBTS and RVPAS groups at the 14-months of age echo. Of these, some patients did not have acceptable echos or not all measures were able to be obtained to calculate the volumes.
Measure: Median (Inter-Quartile Range); unit: ml/m^2.6
Arm/Group | MBTS | RVPAS
Number analyzed (Participants) | 107 | 129
ml/m^2.6 | 83.3 [69.4 to 100.3] | 88.9 [72.6 to 104.7]
Statistical Analysis 1: Comparison: MBTS vs RVPAS; Test type: Superiority or Other; p = 0.07, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Echocardiographic Measures of Heart Size and Function: RV End-systolic Volume Indexed to BSA
Description: Right ventricular end-systolic volume indexed to BSA. Echocardiograms were performed at time points relative to the two palliative surgeries (post-Norwood and pre-Stage II) as well as at the specific time point of 14 months of age.
Time Frame: Measured post-Norwood, an average of 17 days post-Norwood
Population: 241 and 239 patients remained in the MBTS and RVPAS groups at the time of the post-Norwood echo. Of these, some patients did not have acceptable echos or not all measures were able to be obtained to calculate the volumes.
Measure: Median (Inter-Quartile Range); unit: ml/m^2.6
Arm/Group | MBTS | RVPAS
Number analyzed (Participants) | 173 | 194
ml/m^2.6 | 50.1 [40.2 to 61.9] | 44.2 [36.6 to 57.1]
Statistical Analysis 1: Comparison: MBTS vs RVPAS; Test type: Superiority or Other; p = 0.001, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Echocardiographic Measures of Heart Size and Function: RV End-systolic Volume Indexed to BSA
Description: Right ventricular end-systolic volume indexed to BSA^1.3. Echocardiograms were performed at time points relative to the two palliative surgeries (post-Norwood and pre-Stage II) as well as at the specific time point of 14 months of age.
Time Frame: Measured pre-stage II surgery, an average of 15 days pre-stage II surgery
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: ml/m^2.6
Arm/Group | MBTS | RVPAS
Number analyzed (Participants) | 127 | 151
ml/m^2.6 | 63.2 [49.9 to 83.0] | 57.9 [44.6 to 69.9]
Statistical Analysis 1: Comparison: MBTS vs RVPAS; Wilcoxon rank-sum test; Test type: Superiority or Other; p = 0.004, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Echocardiographic Measures of Heart Size and Function: RV End-systolic Volume Indexed to BSA
Description: as for outcome 7
Time Frame: Measured at 14 months of age
Population: as for outcome 5
Measure: Median (Inter-Quartile Range); unit: ml/m^2.6
Arm/Group | MBTS | RVPAS
Number analyzed (Participants) | 107 | 129
ml/m^2.6 | 45.4 [38.5 to 56.6] | 50.5 [39.7 to 60.8]
Statistical Analysis 1: Comparison: MBTS vs RVPAS; Test type: Superiority or Other; p = 0.10, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Echocardiographic Measures of Heart Size and Function: RV Ejection Fraction
Description: Right ventricular ejection fraction: 100 x (RV end-diastolic volume - RV end-systolic volume)/RV end-diastolic volume. Echocardiograms were performed at time points relative to the two palliative surgeries (post-Norwood and pre-Stage II) as well as at the specific time point of 14 months of age.
Time Frame: Measured post-Norwood, an average of 17 days post-Norwood
Population: 241 and 239 patients remained in the MBTS and RVPAS groups at the time of the post-Norwood echo. Of these, some patients did not have acceptable echos or not all measures were able to be obtained to calculate the volumes used to calculate the ejection fraction.
Measure: Mean (Standard Deviation); unit: Percentage of RV end-diastolic volume
Arm/Group | MBTS | RVPAS
Number analyzed (Participants) | 173 | 194
Percentage of RV end-diastolic volume | 44.5 (7.6) | 48.5 (7.6)
Statistical Analysis 1: Comparison: MBTS vs RVPAS; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

10. Secondary Outcome: Echocardiographic Measures of Heart Size and Function: RV Ejection Fraction
Description: as for outcome 9
Time Frame: Measured pre-stage II surgery, an average of 15 days pre-stage II surgery
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Percentage of RV end-diastolic volume
Arm/Group | MBTS | RVPAS
Number analyzed (Participants) | 128 | 151
Percentage of RV end-diastolic volume | 42.9 (7.9) | 44.7 (8.3)
Statistical Analysis 1: Comparison: MBTS vs RVPAS; Test type: Superiority or Other; p = 0.07, t-test, 2 sided

11. Secondary Outcome: Echocardiographic Measures of Heart Size and Function: RV Ejection Fraction
Description: as for outcome 9
Time Frame: Measured at 14 months of age
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: Percentage of RV end-diastolic volume
Arm/Group | MBTS | RVPAS
Number analyzed (Participants) | 107 | 129
Percentage of RV end-diastolic volume | 42.7 (7.4) | 42.7 (8.0)
Statistical Analysis 1: Comparison: MBTS vs RVPAS; Test type: Superiority or Other; p = 0.97, t-test, 2 sided

12. Secondary Outcome: Angiographic Findings: Left Pulmonary Artery Size
Description: Diameter of distal left pulmonary artery. Angiograms were performed at the time points relative to the second palliative surgery (pre-Stage II).
Time Frame: Measured pre-stage II surgery, on average 26 days prior to stage II palliation
Population: These patients had pre-stage II palliation visits with acceptable cardiac catheterizations.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | MBTS | RVPAS
Number analyzed (Participants) | 159 | 191
mm | 5.2 (1.5) | 5.4 (1.7)
Statistical Analysis 1: Comparison: MBTS vs RVPAS; Test type: Superiority or Other; p = 0.54, t-test, 2 sided

13. Secondary Outcome: Angiographic Findings: Right Pulmonary Artery Size
Description: Diameter of distal right pulmonary artery. Angiograms were performed at the time points relative to the second palliative surgery (pre-Stage II).
Time Frame: Measured pre-stage II surgery, on average 26 days prior to stage II palliation
Population: These patients had pre-stage II palliation visits with acceptable cardiac catheterizations.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | MBTS | RVPAS
Number analyzed (Participants) | 159 | 191
mm | 6.1 (2.0) | 5.4 (1.7)
Statistical Analysis 1: Comparison: MBTS vs RVPAS; Test type: Superiority or Other; p < 0.001, t-test, 2 sided

14. Secondary Outcome: Unintended Cardiovascular Interventional Procedures
Description: Unintended cardiovascular procedures included balloon dilation of the shunt or branch pulmonary arteries, stent placement in the shunt or branch pulmonary arteries, shunt revision, crossover between MBTS and RVPAS shunt, balloon dilation, stent placement or surgical revisions of the neo-aorta, and pulmonary artery reconstructions, other than those undertaken as a standard component of the stage II procedure. The number of cardiovascular procedures was analyzed; trial participants may have had more than one unintended cardiovascular. procedure.
Time Frame: From Randomization to 12 months
Measure: Number; unit: procedures
Arm/Group | MBTS | RVPAS
Number analyzed (Participants) | 275 | 274
procedures | 192 | 252
Statistical Analysis 1: Comparison: MBTS vs RVPAS; Test type: Superiority or Other; p = 0.003, Poisson regression; The offset parameter used in the poisson regression was the log of the number of patients in each treatment arm

15. Secondary Outcome: Complications: Total Number Experienced During Norwood Hospitalization
Description: Complications, reported as 'Other Adverse Events' in the safety section, are those adverse events that were not considered serious. Many normal peri-operative occurrences meet the standard criteria of an adverse event; therefore, for this trial a serious adverse event was (a) death, (b) acute shunt failure requiring intervention, (c) cardiac arrest requiring CPR and medications, (d) cardiopulmonary insufficiency requiring ECMO, (e) cardiovascular re-operation (unplanned), (f) necrotizing enterocolitis requiring laparotomy, and (g) any event considered by the study investigator as serious.
Time Frame: Norwood Hospitalization, an average of 36 days
Measure: Number; unit: complications
Arm/Group | MBTS | RVPAS
Number analyzed (Participants) | 275 | 274
complications | 850 | 792
Statistical Analysis 1: Comparison: MBTS vs RVPAS; Test type: Superiority or Other; p = 0.20, Poisson Regression; The offset parameter used in this analysis was the log of the number of patients per treatment arm

16. Secondary Outcome: Complications: Total Number Experienced From Norwood Discharge to Stage II Discharge
Description: as for outcome 15
Time Frame: From Norwood Discharge to Stage II discharge, an average of 4.2 months
Population: These numbers reflect those patients who were discharged from the hospital after the Norwood procedure and were transplant free.
Measure: Number; unit: complications
Arm/Group | MBTS | RVPAS
Number analyzed (Participants) | 219 | 233
complications | 367 | 515
Statistical Analysis 1: Comparison: MBTS vs RVPAS; Test type: Superiority or Other; p = 0.002, Poisson Regression; The offset parameter used in this analysis was the log of the number of patients per treatment arm

17. Secondary Outcome: Complications: Total Number Experienced From Stage II Discharge to 14 Months of Age
Description: as for outcome 15
Time Frame: From Stage II Discharge to 14 Months of Age, an average of 8.9 months
Population: These numbers reflect the number of patients who were discharged from the hospital after the Stage 2 procedure and were transplant-free.
Measure: Number; unit: complications
Arm/Group | MBTS | RVPAS
Number analyzed (Participants) | 176 | 202
complications | 81 | 145
Statistical Analysis 1: Comparison: MBTS vs RVPAS; Test type: Superiority or Other; p = 0.03, Poisson regression; The offset parameter used in this analysis was the log of the number of patients per treatment arm

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the time of randomization through study completion. Adverse events through 12 months after randomization are presented.
Description: Serious Adverse Events: (a) death; (b)acute shunt failure requiring intervention; (c) cardiac arrest requiring CPR and medications; (d) cardiopulmonary insufficiency requiring ECMO; (e) cardiovascular re-operation (unplanned); (f) necrotizing enterocolitis requiring laparotomy; and (g) any other event considered serious by the study investigator.
Arm/Group | MBTS | RVPAS
Serious Adverse Events (participants affected / at risk) | 146/275 | 112/274
Other Adverse Events (participants affected / at risk) | 249/275 | 251/274
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MBTS (N=275) | RVPAS (N=274)
Cardiac arrhythmia (Cardiac disorders) | 7 (8) | 9 (10)
Cardiac general (Cardiac disorders) | 97 (111) | 63 (73)
Coagulation (Blood and lymphatic system disorders) | 1 (1) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 3 (3) | 3 (3)
Hemorrhage/bleeding (Blood and lymphatic system disorders) | 4 (4) | 6 (6)
Infection (Infections and infestations) | 7 (7) | 9 (9)
Metabolic/laboratory (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Musculoskeletal/soft tissue (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neurology (Nervous system disorders) | 5 (6) | 4 (4)
Pulmonary/upper respiratory (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 11 (11)
Renal/genitourinary (Renal and urinary disorders) | 3 (3) | 3 (3)
Surgery/intra-operative injury (Surgical and medical procedures) | 4 (4) | 4 (4)
Vascular (Vascular disorders) | 35 (36) | 29 (29)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MBTS (N=275) | RVPAS (N=274)
Cardiac disorders (Cardiac disorders) | 161 (316) | 148 (266)
Gastrointestinal (Gastrointestinal disorders) | 93 (138) | 94 (133)
Hematologic (Blood and lymphatic system disorders) | 48 (64) | 57 (73)
Infectious (Infections and infestations) | 156 (313) | 172 (401)
Neurological (Nervous system disorders) | 35 (51) | 53 (77)
Respiratory (Respiratory, thoracic and mediastinal disorders) | 154 (285) | 172 (387)
Renal (Renal and urinary disorders) | 39 (41) | 27 (28)
Vascular (Vascular disorders) | 32 (34) | 34 (38)

LIMITATIONS AND CAVEATS:
As in all surgical trials comparing two operations, it was not possible to blind the personnel caring for the subjects to the intervention. However, the components of the primary endpoint, death and transplantation, are discrete objective events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No